CLINICAL TRIAL: NCT06200727
Title: Application of Platelet-rich Fibrin(PRF) Membrane in Ophthalmic Diseases
Brief Title: Platelet-rich Fibrin(PRF) Membrane in Ophthalmic Diseases
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Lei Du (Other)
Responsible Party: Sponsor-Investigator, Lei Du, deputy chief physician, Renmin Hospital of Wuhan University
Organization: Renmin Hospital of Wuhan University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WDRY2022-K197
Record Dates: First submitted 2023-12-11; First posted 2024-01-11 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2024-01

CONDITIONS: Platelet-rich Fibrin; Macular Holes; Pterygium; Glaucoma
Keywords: PRF; pterygium; macular hole; corneal ulcer
MeSH Terms: conditions — Retinal Perforations; Pterygium; Glaucoma; Corneal Ulcer | interventions — Trabeculectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- PRF membrane in macular hole (Experimental): To observe the healing and visual recovery of a macular hole, the macular hole was filled with a PRF membrane. Before the participant went into the operating theatre, a blood sample was taken from the anterior elbow vein using a 5 ml tube without anticoagulants. The middle layer of blood after centrifugation was PRF. After retrobulbar anesthesia and removal of the posterior vitreous cortex. In the PRF group, PRF membrane was utilized to fill the macular hole after the ILM was peeled. Then the eyeball was filled with sterile air after adequate air-liquid exchange. At the end of the operation, tobramycin dexamethasone ophthalmic ointment was applied to the operated eye with pressure, and the participant was instructed to maintain a prone position for 7 days after the operation.
  Interventions: Procedure: PRF membrane tamponade surgery in macular hole
- Internal limmiting membrane(ILM) peeling in macular hole (Active Comparator): After retrobulbar anesthesia and removal of the posterior vitreous cortex, the control group underwent the procedure of peeling the ILM. The ILM was completely removed from the retina. Then the eyeballs were filled with sterile air after adequate air-liquid exchange.
  At the end of the operation, tobramycin dexamethasone ophthalmic ointment was applied to the operated eye with pressure, and the participant was instructed to maintain a prone position for 7 days after the operation.
  Interventions: Procedure: ILM peeling in macular hole
- PRF membrane transplantation in pterygium (Experimental): Following the removal of the pterygium, the prepared PRF was cut to match the size of the exposed scleral surface. It was then placed on the sclera and secured to the surrounding conjunctiva using 3-7 interrupted sutures of 10-0 nylon thread. This was done to ensure that the PRF implant was perfectly aligned with the conjunctiva.
  Interventions: Procedure: PRF membrane grafting in pterygium
- Autologous conjunctival transplantation in pterygium (Active Comparator): After the pterygium removal surgery, to restore the eye, participants need to undergo a corneal limbal stem cell transplant. The transplanted stem cells should be the same size as the exposed scleral surface above the temporal part of the eye. When transferring the transplant, ensured that the corneal edge of the grafted conjunctival flap was positioned opposite to the cornea. Closed the flap to the peripheral conjunctiva with 3-7 interrupted sutures using 10-0 nylon thread. Fixed the conjunctival flap to the surrounding conjunctiva with sutures, and covered the sclera with the surrounding bulbar conjunctiva.
  Interventions: Procedure: Autologous conjunctival transplantation in pterygium
- PRF membrane transplantation in trabeculectomy for glaucoma (Experimental): The surgical procedure involved the creation of a scleral flap and conjunctiva in the usual manner. The subflap tissue was rinsed with balanced saline and then a small piece of tissue (measuring 1.5mm x 2mm) was removed from the inferior trabecular tissue of the scleral flap. In the corresponding position, peripheral iris excision was performed and the iris was rinsed to remove lost pigment in the vicinity of the incision. Once the orientation was verified, the PRF membrane was placed under the scleral flap.
  Interventions: Procedure: autologous PRF membrane grafting in trabeculectomy for glaucoma
- Amniotic membrane in trabeculectomy for glaucoma (Active Comparator): The surgical procedure began with creating the scleral flap and conjunctiva in the usual manner. The sub flap tissue was then rinsed with balanced saline, and a piece of tissue measuring 1.5mm x 2mm was excised from the inferior trabecular tissue of the scleral flap. Next, peripheral iris excision was performed in the corresponding position and the iris was rinsed to remove pigment in the vicinity of the incision. To control the tension of the sutures, the amniotic membrane was placed under the scleral flap, followed by meticulous suturing of the conjunctival flap.
  Interventions: Procedure: Amniotic membrane in trabeculectomy for glaucoma
- PRF membrane transplantation in corneal ulcer (Experimental): The necrotic tissue of the corneal ulcer was cleared to expose the local fresh tissue, and the PRF group prepared PRF membrane and covered the surface of the test eye, and the autologous PRF membrane was continuously sutured to the corresponding surrounding tissues using 10-0 absorbable sutures so that the PRF membrane covered the entire portion of the lesion and was able to be anchored to it.
  Interventions: Procedure: PRF membrane grafting incorneal ulcer
- Amniotic membrane in corneal ulcer (Active Comparator): The necrotic tissue of the corneal ulcer was removed to reveal the fresh tissue in the area. After that, the excess amniotic membrane was carefully extracted and placed over the affected eye's surface. The membrane was then attached securely to the surrounding tissue using 10-0 absorbable sutures, covering the entire lesion and holding it in place for proper healing.
  Interventions: Procedure: Amniotic membrane in corneal ulcer

INTERVENTIONS:
Procedure: PRF membrane tamponade surgery in macular hole — A specially formulated PRF membrane, as described previously, was filled into the macular hole to promote fissure repair.
  Arms: PRF membrane in macular hole
Procedure: ILM peeling in macular hole — The treatment of the macular hole was ILM peeling.
  Arms: Internal limmiting membrane(ILM) peeling in macular hole
Procedure: PRF membrane grafting in pterygium — Used of autologous PRF membrane to cover the exposed conjunctiva after pterygium excision.
  Arms: PRF membrane transplantation in pterygium
Procedure: Autologous conjunctival transplantation in pterygium — Used of autologous conjunctiva to cover exposed sclera after pterygium excision
  Arms: Autologous conjunctival transplantation in pterygium
Procedure: autologous PRF membrane grafting in trabeculectomy for glaucoma — Used of autologous PRF membranes to cover the exposed sclera after trabeculectomy for glaucoma.
  Arms: PRF membrane transplantation in trabeculectomy for glaucoma
Procedure: Amniotic membrane in trabeculectomy for glaucoma — Used of amniotic to cover the exposed sclera after trabeculectomy for glaucoma.
  Arms: Amniotic membrane in trabeculectomy for glaucoma
Procedure: PRF membrane grafting incorneal ulcer — After surgical debridement of corneal ulcers, autologous PRF membrane was placed over the corneal wound to promote corneal healing
  Arms: PRF membrane transplantation in corneal ulcer
Procedure: Amniotic membrane in corneal ulcer — After surgical debridement of corneal ulcers, autologous amniotic membrane was placed over the corneal wound to promote corneal healing
  Arms: Amniotic membrane in corneal ulcer

SUMMARY:
The goal of this clinical trial is to observe the role of PRF in treating ophthalmic diseases.The efficacy and safety of PRF were validated for four ophthalmic conditions: macular hole, pterygium, corneal ulcer, and patients undergoing trabeculectomy for glaucoma. The main question aims to answer is PRF's effectiveness in ocular surface and fundus diseases. Participants will be divided into 2 groups, the experimental group will be treated with PRF and the control group will be treated with conventional surgery, with a 12-month postoperative follow-up to determine the role of PRF on wound healing in ophthalmic diseases.

DETAILED DESCRIPTION:
Patients suffering from pterygium, macular hole, corneal ulcer, and glaucoma requiring for trabeculectomy , who visited Renmin Hospital of Whuhan University, were chosen to participate in this study. The participants were randomly divided into the experimental group (PRF group) and the control group (conventional group). The PRF group received PRF membrane treatment, while the conventional group received conventional surgical treatment. Before and after surgery, participants underwent a comprehensive ophthalmological exam at 1 week, 1 month, 3 months, 6 months, and 12 months.

The outcome indicators are monitored and can vary depending on the disease. Participants with pterygium were examined for graft dissolution and complications. Participants with macular hole were monitored for hole closure, visual acuity recovery, and retinal blood flow recovery. Participants with corneal ulcer were monitored for lesion healing and complications such as degree of corneal vascularization and opacity. Participants with glaucoma were monitored for postoperative intraocular pressure (IOP), degree of conjunctival leakage in the filtration zone, and degree of scarring in the filtration zone.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of macular hole confirmed by fundus examination;
2. Diagnosis of pterygium by slit lamp;
3. Patients requiring trabeculectomy for glaucoma;
4. Diagnosis of corneal ulcer confirmed by slit lamp.

Exclusion Criteria:

1. Combination of other active ophthalmic diseases, such as acute conjunctivitis and uveitis;
2. Previous history of ophthalmic trauma and ophthalmic surgery;
3. Recent use of anticoagulant or antiplatelet drugs;
4. Combination of serious systemic diseases such as hypertension and diabetes mellitus.

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Whether the macular hole is closed in participants with macular hole(Unit: yes/no) | Pre-operation, and at 1 week, 1 month, 3 months, and 6 months post-operation.
  Using optical coherence tomography（OCT ）to see if the macular hole is healing to compare the healing rate between the PRF membrane filling group and the ILM peeling group.
Whether the wound heals completely after pterygium excision in participants with pterygium(Unit: yes/no) | Pre-operation, and at 1 week, 1 month, 3 months, and 6 months post-operation.
  Observation of the anterior segment of the eye using a slit lamp to determine whether the wound is healed after pterygium excision and to compare the healing rate between the PRF membrane-covered group and the autologous conjunctival-covered group.
IOP in participants undergoing trabeculectomy for glaucoma(Unit: mmHg) | Pre-operation, and at 1 week, 1 month, 3 months, and 6 months post-operation.
  Measurement of IOP using an IOP meter to compare the effect of IOP reduction in glaucoma treatment in the PRF membrane group and the amniotic membrane group.
Whether the corneal ulcer is healing in participants with corneal ulcer(Unit: yes/no) | Pre-operation, and at 1 week, 1 month, 3 months, and 6 months post-operation.
  The investigators use a slit lamp to examine the anterior segment of the eye to assess the corneal wound healing rate. The PRF membrane-covered group is compared to the control group.

SECONDARY OUTCOMES:
Best-corrected visual acuity (BCVA) in participants with macular hole(Unit: logMAR) | Pre-operation, and at 1 week, 1 month, 3 months, and 6 months post-operation.
  Measurement of BCVA in participants with macular holes using an international standard logarithmic visual acuity chart.
Occurrence of complications in participants with pterygium(Unit: rate) | Pre-operation, and at 1 week, 1 month, 3 months, and 6 months post-operation.
  Using a slit lamp, visualizing the anterior eye segment to detect complications in participants with pterygium.
Degree of tissue scarification in participants undergoing trabeculectomy for glaucoma(Unit: mild, moderate, severe) | Pre-operation, and at 1 week, 1 month, 3 months, and 6 months post-operation.
  Viewing the anterior segment of the eye using a slit lamp to determine the extent of tissue scarring in participants undergoing trabeculectomy for glaucoma.
Occurrence of complications in participants with corneal ulcer(Unit: rate) | Pre-operation, and at 1 week, 1 month, 3 months, and 6 months post-operation.
  Using a slit lamp, visualizing the anterior eye segment to detect complications in participants with corneal ulcer.

CONTACTS AND LOCATIONS:
Overall Officials: Lei Du, Principal Investigator — Renmin Hospital of Wuhan University
Locations (1):
- Eye Center, Renmin Hospital of Wuhan University, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No
This is a new technology and the information may be of commercial value to healthcare organisations and pharmaceutical companies. If this data is made public, it may result in other organisations or businesses gaining access to this information, which may affect the organisation's competitive advantage.

REFERENCES:
- [Background] Yang N, Xing Y, Zhao Q, Zeng S, Yang J, Du L. Application of platelet-rich fibrin grafts following pterygium excision. Int J Clin Pract. 2021 Oct;75(10):e14560. doi: 10.1111/ijcp.14560. Epub 2021 Jul 5. PMID 34155746
- [Result] Yang N, Zeng S, Yang J, Lu G, Du L. Application of Platelet-Rich Fibrin Transplantation for Large Macular Hole. Curr Eye Res. 2022 May;47(5):770-776. doi: 10.1080/02713683.2022.2029906. Epub 2022 Mar 22. PMID 35179414
- [Derived] Lu G, Zeng S, Huang R, Du L. Platelet-rich Fibrin Membrane Transplantation for the Treatment of Highly Myopic Macular Hole Retinal Detachment. Ophthalmol Ther. 2024 Sep;13(9):2425-2443. doi: 10.1007/s40123-024-00997-w. Epub 2024 Jul 26. PMID 39060701